CLINICAL TRIAL: NCT01163812
Title: A Phase-II Clinical Trial of Laparoscopy-Assisted Distal Gastrectomy With D2 Lymph Node Dissection for Gastric Cancer
Brief Title: Clinical Trial for Laparoscopic D2 Gastrectomy
Acronym: NCC181
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Young-Woo Kim/ head, National Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-2005181
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Last update posted 2010-07-19 (Estimated); Status verified 2010-07

CONDITIONS: Gastric Cancer
Keywords: D2 lymph node dissection
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laparoscopic D2 gastrectomy (Experimental)
  Interventions: Procedure: Laparoscopic D2 distal gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic D2 distal gastrectomy — Under general endotracheal anesthesia, Five or six ports are used. Lymph node dissection and ligation of vessels are carried out in the laparoscopic field. A partial omentectomy encompassing perigastric nodes is performed laparoscopically. D2 lymphadenectomy is carried out according to the guidelines of the "The Japanese Research Society for Gastric Cancer" for the corresponding location of the primary tumor. A 5- to 6-cm small incision is made transversely in RUQ of the abdomen. Through the incisional window, the stomach is removed from the abdominal cavity and resected. A Billroth-I gastroduodenostomy using an EEA stapler and GIA or a Billroth-II gastrojejunostomy with a hand-sewing technique is performed. The abdomen is then closed after hemostasis is achieved.
  Other Names: LADG

SUMMARY:
Objectives of this study was to determine whether laparoscopy-assisted distal gastrectomy (LADG) with complete D2 lymph node dissection for gastric cancer is a safe and effective surgical option.

Methods: total 64 patients, who are diagnosed preoperatively as having T1-2, N0-1 or M0 gastric cancer, will be prospectively enrolled to undergo LADG with D2 lymph node dissection; two surgeons with experience of over 50 cases of laparoscopic gastrectomy performed the procedures. The compliance rate, defined as cases with no more than one missing lymph node station according to the Japanese Research Society of Gastric Cancer (JRSGC) lymph node grouping, for the open gastrectomy with D2 lymph node dissection was 66.0% in a pilot study and was used for calculations of sample size. Compliance rate and other surgical outcomes, including the number of retrieved lymph nodes from each lymph node station, morbidities, mortalities and conversion rate will be analyzed.

DETAILED DESCRIPTION:
Gastric cancer is the most common cancer in Korea; the overall age-standardized incidence rates of gastric cancer in Korea have been reported to be 69.6 per 100,000 among males and 26.8 per 100,000 among females in 2000.

Treatment modalities for resectable gastric cancer include endoscopic mucosal resection (EMR), laparoscopy-assisted gastrectomy (LAG) and conventional open gastrectomy. Laparoscopic cancer surgery has been reported to be an acceptable alternative to open surgery in patients with colorectal cancer. However, in gastric cancer, laparoscopic surgery has not yet been validated and, thus, is performed only in a limited number of patients with early gastric cancer; this is due to the technical difficulty in systematic lymph node dissection. For the treatment of advanced gastric cancer (AGC), in countries including Korea and Japan, gastrectomy with D2 lymph node dissection has been the standard operation. With the recent progress in diagnostic techniques, accumulation of experience with laparoscopy-assisted distal gastrectomy (LADG) for early gastric cancer and the increasing interest in a better quality of life, there has been an effort to apply minimally invasive techniques to the treatment of AGC. However, there has been no clinical trial to test the oncological feasibility of LADG with D2 lymph node dissection. There is only one phase-II study that evaluated whether the morbidity associated with LADG was higher than that of open gastrectomy.

Before the indications for LADG can be extended to include patients with advanced cancer, the status of surgical expertise for complete D2 lymph node dissection requires investigation using a prospective clinical study design. If this approach is shown to be feasible, a randomized prospective clinical trial, to compare survival and other surgical outcomes, would be the next step in validating this technique for this group of patients.

This study is to be performed according to the Helsinki Declaration. The study was approved by the Ethics Subcommittee at the National Cancer Center for Research Involving Human Subjects (no. NCCCTS-2005181). All patients will be provided written informed consent before entering the study.

Sample size The sample size was based on the alpha error at 0.05 and 90% of power and the accepted margin of the difference in the compliance rate at 10% based on a non-inferiority test. The target was chosen from the primary end point of the study. For the patients who underwent LADG with D2 lymph node dissection, the compliance rate-defined as cases in which there was no more than one missing lymph node station according to the guidelines of "The Japanese Research Society for Gastric Cancer" (JRSGC) lymph node grouping,11,12-was set up to 55%; for the patients with open distal gastrectomy with D2 lymph node dissection, it was 66%, based on a pilot study. We performed a pilot study to determine the compliance rate in 100 cases of open distal gastrectomy with D2 lymph node dissection before enrollment started. When the data was used for the formula, the total sample size required was determined to be 60 patients. When we added 10% for expected follow-up loss, the total sample size was calculated to be 66 patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the stomach,
* Age between 18 and 75 years, performance status of ECOG 0-1
* Signed informed consent
* Location of the primary tumor in the antrum, angle and lower body
* No evidence of distant metastasis or invasion to adjacent organs or serosal infiltration,
* Enlarged lymph node size 2 cm or less on CT and no conglomerate nodes or regional
* Lymph node metastasis confined to perigastric nodes (N1) as shown on by CT and EUS

Exclusion Criteria:

* Metastatic disease, previous history of malignancy in any organ, any co-morbidity
* Obviating major surgery, contraindication to laparoscopy such as severe cardiac disease
* Abdominal wall hernias, diaphragmatic hernias, uncorrected coagulopathies, portal hypertension, pregnancy, previous upper abdominal surgery, complicated cases requiring emergency surgery, and an accompanying surgical condition requiring surgery at the same time

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2006-04; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Compliance of lymph node dissection | immediate postoperative 1 week
  noncompliance : if two or more nodal station is vacant, it is a noncompliant D2 gastrectomy.

SECONDARY OUTCOMES:
Proportion of patients with retrieved lymph nodes less than 26 | Postoperative 1 week
operative complications | Postoperative 1 month
  intra, and postopertive complications related to operation.
operative time | postoperative 1 day
estimated blood loss | postoperative 1 day
  blood loss during operation.
amount of administered analgesics | Postoperative 1 week
time to diet | postoperative 1 week
time to return of bowel movement | postoperative 1 week
hospital stay | postoperative 1 week
distance to resection margin and number of harvested lymph nodes | postoperative 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Young-Woo Kim, MD, PhD, Principal Investigator — NCC Korea
Locations (1):
- National Cancer Center, Goyang, Gyeonggido, South Korea

REFERENCES:
- [Background] Ryu KW, Kim YW, Lee JH, Nam BH, Kook MC, Choi IJ, Bae JM. Surgical complications and the risk factors of laparoscopy-assisted distal gastrectomy in early gastric cancer. Ann Surg Oncol. 2008 Jun;15(6):1625-31. doi: 10.1245/s10434-008-9845-x. Epub 2008 Mar 14. PMID 18340493
- [Result] Lee JH, Kim YW, Ryu KW, Lee JR, Kim CG, Choi IJ, Kook MC, Nam BH, Bae JM. A phase-II clinical trial of laparoscopy-assisted distal gastrectomy with D2 lymph node dissection for gastric cancer patients. Ann Surg Oncol. 2007 Nov;14(11):3148-53. doi: 10.1245/s10434-007-9446-0. Epub 2007 Aug 20. PMID 17705092
- [Result] Lee SE, Kim YW, Lee JH, Ryu KW, Cho SJ, Lee JY, Kim CG, Choi IJ, Kook MC, Nam BH, Park SR, Kim MJ, Lee JS. Developing an institutional protocol guideline for laparoscopy-assisted distal gastrectomy. Ann Surg Oncol. 2009 Aug;16(8):2231-6. doi: 10.1245/s10434-009-0490-9. Epub 2009 May 9. PMID 19430842